CLINICAL TRIAL: NCT02692846
Title: Williams Syndrome Skin and Vascular Elasticity Study (WS-SAVE Study)
Brief Title: WS-SAVE Study (Williams Syndrome Skin and Vessel Elasticity Study)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160063; 16-H-0063
Record Dates: First submitted 2016-02-25; First posted 2016-02-26 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-05-05

CONDITIONS: Williams Syndrome; Cardiovascular Disease; Multisystem Developmental Disorder; Elastin Gene Deletion; Hypertension
Keywords: CONNECTIVE TISSUE DISEASES; Cardiovascular Disease; Elastin Gene Mutation; Multisystem Developmental Disorder; Natural History
MeSH Terms: conditions — Williams Syndrome; Cardiovascular Diseases; Hypertension; Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control participants with connective tissue disease: Not have a diagnosis of WS. Have a clinical or molecular diagnosis of connective tissue disease, between the ages of 1 and 70 years old
- Unaffected Control participants: Not have a diagnosis of WS or other connective tissue disease, between the ages of 1 and 70 years old
- WS participants: Have diagnosis of WS, between the ages of 5 and 70 years old. Be able to tolerate blood pressure measurements.

SUMMARY:
Background:

Williams Syndrome (WS) is a genetic disorder. People with WS have less of a protein that allows parts of the body to stretch than other individuals. Researchers are interested in the stretchiness of the skin of people with WS and how it may relate to cardiovascular problems some people with WS develop. They are also interested in identifying exposures such as medications that may change the elasticity of the skin and vessels.

Objective:

To learn more about the skin and blood vessels in individuals with WS and how those tissues change over time.

Eligibility:

People ages 5-70 with WS.

People ages 1-70 with a medical condition that affects connective tissue.

Design:

Participants will be screened with a review of their medical records.

Participants will have 1 visit. Participants with WS may do so at a Williams Syndrome Association family meeting or camp, or at NIH. Other participants will be seen at NIH.

During the visit, participants will have height, weight, and blood pressure measured.

Researchers will listen to the participant s chest and abdomen.

Participants skin will be examined. It may be photographed.

Participants will have photos of their eyes and face taken.

Researchers will use a DermaLab Suction Cup Probe. A small suction cup will be placed on the arm with a sticker. It will pull lightly on the skin. This allows a computer to measure skin flexibility.

Researchers will use a SphygmoCor. A probe that looks like a dull pencil will be placed on the wrist, neck, and groin area. A computer will measure how fast the pulse is moving and will estimate blood vessel flexibility.

Participants may be invited to have these procedures repeated at a later date (2 years from now or more).

DETAILED DESCRIPTION:
Williams syndrome (WS) is a multisystem developmental disorder caused by deletion of 26-28 genes, including the elastin gene, located on chromosome 7q11.23. Cardiovascular disease in WS, including obstructive vascular disease and hypertension, and relatively mild skin changes are caused by the elastin gene deletion. Even though all WS subjects are missing one copy of this gene, the expression of cardiovascular problems is highly variable, ranging from no significant disease to severe generalized arteriopathy leading to infant death. The causes of vascular variability are currently unknown, and male gender is the only disease modifier described to date. Clinically, skin is described as abnormally soft, smooth and easily mobilized , while ultrastructurally the elastic fibers are abnormal with reduced amorphous elastin.

The overall objective of this study is to establish quantitative norms that can be used to determine the severity of vascular disease in elastin insufficiency and then to identify risk factors that contribute to that variability. It is also important to determine how stable/variable these findings are over time.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

For WS participants:

Individuals participating in this study must:

* Have a diagnosis of WS
* Be between the ages of 5 and 70 years old
* Be able to tolerate blood pressure measurements
* Have a parent/guardian available to provide consent and assist in answering medical questions.
* Express willingness to schedule an in-person assessment with us.

The only indication for study staff to terminate an individual s participation in this study would be if the family is unable to schedule an in-person assessment with us.

For unaffected control participants:

Individuals participating in this study must:

* Not have a diagnosis of WS or other connective tissue disease.
* Be between the ages of 1 and 70 years old
* If a minor, have a parent/guardian available to provide consent and assist in answering medical questions.

For control participants with connective tissue disease:

Individuals participating in this study must:

* Not have a diagnosis of WS
* Have a clinical or molecular diagnosis of connective tissue disease.
* Be between the ages of 1 and 70 years old
* If a minor, have a parent/guardian available to provide consent and assist in answering medical questions.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit three subject populations, individuals with WS and two control populations, one unaffected and one with known connective tissue disease. Affected subjects being screened for a research protocol or already on a research protocol at the NIH Clinical Center (CC) may be contacted by their physician about this study.@@@Subjects who are able to visit the NIH CC will be enrolled in person by the PI or approved AIs of the study, as mentioned in the previous section. For off-site subjects, the PI or approved AIs of this protocol may conduct an in-person, off-site meeting with the subject to carefully explain the research objectives, procedure(s), and relevant risks and discomforts of this protocol or attend WSA meetings that occur every 2 years and consent the subject at the meeting place.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
To identify risk factors that contribute to the variability in cardiovascular and skin phenotype in individuals with Williams syndrome, primarily focusing on differences in elasticity and compliance | 2-4
  1) clinical and objective assessment of the vasculature and skin in individuals with WS, focusing on its elasticity; 2) analysis as to whether skin and vascular elasticity correlate with each other. 3) identification of genetic risk factors contributing to their variability, and 4) non-invasive measurement of urine biomarkers for oxidative stress. Note: with the NHLBI initial submission, items # 3 and 4 above will no longer be evaluated.

SECONDARY OUTCOMES:
To determine how stable/variable these findings are over time | 2-4 years
  Skin and vascular elasticity analysis may be repeated in willing individuals at later dates (at least 2 years apart) to assess changes in the measurements with time.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Boehm, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pober BR. Williams-Beuren syndrome. N Engl J Med. 2010 Jan 21;362(3):239-52. doi: 10.1056/NEJMra0903074. No abstract available. PMID 20089974
- [Background] Urban Z, Peyrol S, Plauchu H, Zabot MT, Lebwohl M, Schilling K, Green M, Boyd CD, Csiszar K. Elastin gene deletions in Williams syndrome patients result in altered deposition of elastic fibers in skin and a subclinical dermal phenotype. Pediatr Dermatol. 2000 Jan-Feb;17(1):12-20. doi: 10.1046/j.1525-1470.2000.01703.x. PMID 10720981
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-H-0063.html